CLINICAL TRIAL: NCT05108701
Title: Individual Mindfulness-Based Cognitive Therapy vs. Cognitive Behavior Therapy and Treatment As Usual as Treatment for Major Depressive Disorder: A Pilot Study.
Brief Title: Individual MBCT vs. CBT in Major Depression: A Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G6302357
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Parallel, two-arm, randomised pilot trial comparing Individual MBCT with Individual CBT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-MBCT (Experimental): Participants randomized to I-MBCT (Mindfulness-Based Cognitive Therapy) receive 12 weekly 60- minute sessions of I-MBCT according to the protocol of Segal et al. (2002), integrated with the "theme, rationale, intention and practice" skills (TRIP) protocol (Woods et al. 2016, 2019). The original MBCT protocol, created for eight group sessions lasting two hours, is adapted to twelve individual sessions.
  Interventions: Behavioral: Individual Psychotherapy
- CBT (Active Comparator): Participants randomized to Individual Cognitive Behavioural Therapy (CBT) receive 12 weekly 60-minute individual sessions of standard CBT strategies following Beck et al. (1979). Participants receive a copy of Greenberger and Padesky's Mind over Mood (The Guilford Press, 1995) for use during the intervention.
  Interventions: Behavioral: Individual Psychotherapy

INTERVENTIONS:
Behavioral: Individual Psychotherapy — Psychotherapy using meditation, yoga, through being in the present moment a non judgmental way and open minded

SUMMARY:
Background: Depression is a highly recurrent disorder, which often requires lifelong treatment. Psychotherapy has an important role in the treatment of depression, both in the treatment of the acute phase and in prevention of relapses. Mindfulness-based therapies have become popular in the last decade. Mindfulness-based Cognitive Therapy (MBCT) is an established treatment for relapse prevention in Major Depressive Disorder (MDD) and there is preliminary evidence of its efficacy in treating acute symptoms. Several studies have highlighted the benefits of MBCT in reducing the severity of depressive symptoms in patients diagnosed with a current Major Depressive Episode, as indicated by some meta-analyses showing that MBCT is more effective than treatment as usual in decreasing depressive symptoms and equivalent to active treatments. However, the results at follow-up were less conclusive, due to the limited number of studies and moderate-to-large heterogeneity within the subgroups.

A number of studies have examined the effects of MBCT on a larger spectrum of factors that can affect the severity of depression. In patients with MDD, MBCT was more effective than treatment as usual in decreasing rumination, worry, negative affect and dysfunctional attitudes, increasing mindfulness skills and positive affect and improving sleep and quality of life. However, data comparing the specific effect of MBCT with other active treatments (for example Cognitive Behavioural Therapy, CBT) are lacking.

Most trials exploring the efficacy of MBCT have been conducted with group MBCT, but there is less evidence about the use of individual MBCT (I-MBCT). Individual MBCT may have some advantages, compared with group therapy, such as better attendance and higher efficacy in major depression, when compared with group therapy. Furthermore, the individual format can often be better tailored to a specific patient, with a slower progression and a longer number of sessions, if needed.

Objective: The primary objective of this pilot trial was to test the feasibility of a larger randomized trial examining the changes in depressive and anxiety symptoms, rumination, mindfulness, emotion regulation, behavioral activation and negative automatic thoughts during I-MBCT and cognitive behavioural therapy (CBT). Further objectives were: (a) replicating studies evaluating the efficacy of I-MBCT to improve depression, in particularly in patients diagnosed with a major depressive disorder; (b) assessing the persistence of benefits of I-MBCT after the end of treatment; (c) comparing the effects of I-MBCT with CBT, not only on depressive symptoms, but also on factors which are specifically targeted by MBCT, such as rumination and mindfulness; explore possible predictors of outcome of MBCT.

Hypotheses: We make the following hypotheses: a) a larger trial comparing I-MBCT with CBT examining the changes of depressive and anxiety symptoms, rumination, mindfulness, emotion regulation, behavioral activation and negative automatic thoughts is feasible, with recruitment rates and drop-off rates consistent with those usually observed among participants with current major depression; b) the levels of depressive and anxiety symptoms, rumination, emotion dysregulation, and negative automatic thoughts will decrease during I-MBCT, while the levels of mindfulness and behavioral activation will increase, with effect sizes similar to those observed in CBT; c) the changes in depressive and anxiety symptoms, rumination, emotion dysregulation, negative automatic thoughts, mindfulness and behavioral activation will be maintained at follow-up; d) the changes in mindfulness and rumination dimensions are expected to be larger during MBCT than CBT; these analyses will be exploratory, given the state of knowledge; d) we will explore the role of predictors of clinical variables, such as earlier age at onset of the mood disorder; longer and more severe current episode; presence of current comorbidity with anxiety disorders, initial levels of anxiety, behavioral activation, emotion dysregulation and of the history of severe childhood maltreatment in predicting the outcome to MBCT and CBT.

DETAILED DESCRIPTION:
The trial is a parallel, two-arm, randomised pilot trial (Ottawa, Ontario, Canada). Participants will be recruited from the Mood and Anxiety Program of the Royal Ottawa Mental Health Centre, which is a specialized tertiary care centre, and from two psychiatrists working in community.

Procedure Participants will be referred to the study by the treating psychiatrist, then screened in a telephone interview by the research coordinator; the eligibility criteria will be finally assessed by a psychiatrist involved in the study and by the research coordinator. The psychiatrist will administer the Structured Clinical Interview (SCID) for DSM-IV-TR (First et al. 2002) and collect the information related to clinical variables: previous hospitalizations, history of suicide attempts, comorbidity with a current anxiety disorder, age at onset of the mood disorder, number of previous major depressive episodes, duration of the current episode, severity of the current depressive episode, use of alcohol or street drugs, family history of affective disorders, and number of chronic medical conditions. The research coordinator will assess the severity of depression using the HAMD-17. If the criteria of eligibility to the study were satisfied, participants will be asked to sign an informed written consent. Individuals meeting study criteria will be randomly assigned by computer-generated numbers to treatment with either I-MBCT or CBT (1:1). Participants included in the trial will be followed by the referring clinician. Concurrent use of psychotropics will be allowed. Concomitant treatment with any form of structured "bona fide" psychotherapy is not permitted during the study.

Participants randomized to I-MBCT receive 12 weekly 60- minute sessions of I-MBCT according to the protocol of Segal et al. (2002), integrated with the "theme, rationale, intention and practice" skills (TRIP) protocol (Woods et al. 2016, 2019). The original MBCT protocol, created for eight group sessions lasting two hours, is adapted to twelve individual sessions.

Participants randomized to CBT receive 12 weekly 60-minute individual sessions of standard CBT strategies following Beck et al. (1979). Participants receive a copy of Greenberger and Padesky's Mind over Mood (The Guilford Press, 1995) for use during the intervention.

Data Analyses The statistical analysis will be performed on the overall sample of patients who will start the treatment. As this was a feasibility study, a formal sample size calculation was not required. We applied the "rule of thumb" recommended by Julious (2005), suggesting a minimum of 12 participants per treatment arm, which optimizes the gain in precision around the mean. Pre-treatment demographic and clinical characteristics will be compared between I-MBCT and CBT treatment using univariate analyses (t-test for continuous variables and Fisher test for categorical variables).

The primary outcome will be the HAM-D. The changes in depressive and anxiety symptoms, rumination, emotion dysregulation, and negative automatic thoughts during MBCT and at follow-up will be tested through linear mixed-effects models (LMM, SPSS Mixed procedure). Interaction between time and treatment will be use to compare the changes during MBCT and CBT. Multiple regression analyses will be used to test the value of clinical variables in predicting the changes in severity of depressive symptoms during psychotherapy, adjusting for age, gender and baseline depressive severity .

To evaluate the strength of the changes in outcome variables (depressive and anxiety symptoms, rumination, emotion dysregulation, and negative automatic thoughts) during I-MBCT and CBT, within-group effect sizes of the change pre- and post-treatment using Cohen's delta for repeated measures will be used.

ELIGIBILITY:
Inclusion Criteria: a) Diagnosis of MDD, current episode mild to moderate or in partial remission, according to the Diagnostic and Statistical Manual of Mental Disorders - DSM-IV criteria; b) Hamilton rating scale for Depression (HAMD-17), total score between 8 and 18, included; c) age between 18 and 65 years, d) able to comply with the study protocol, e.g. able to attend weekly sessions; and e) English speaking and able to provide informed consent.

Exclusion Criteria: a) a current diagnosis of bipolar disorder, substance use disorder, schizophrenia or primary personality disorder; b) a trial of electroconvulsive therapy (ECT) in the past 6 months; c) depression secondary to a concurrent medical disorder; d) current practice of meditation more than once per week or yoga more than twice per week; and e) treated with MBCT or CBT in the previous year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Hamilton for Depression - 17 items | 10 minutes
  clinician-rated scale measure of depression severity

SECONDARY OUTCOMES:
Beck Depression Inventory - Depression | 3 minutes
  self-rated measure of depression severity
Five Facet Mindfulness Questionnaire | 3 minutes
  self-rated measure of mindfulness
Reflection Rumination Questionnaire - Rumination subscale (RRQ) | 3 minutes
  self-rated measure of rumination
Difficulties in Emotion Regulation Scale | 3 minutes
  self-rated measure of emotion regulation
Automatic Thoughts Questionnaire | 3 minutes
  self-rated measure of negative automatic thoughts
Beck Anxiety Inventory | 3 minutes
  self-rated measure of anxiety
Behavioral Activation for Depression Scale | 3 minutes
  self-rated measure of behavioural activation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tovote KA, Fleer J, Snippe E, Peeters AC, Emmelkamp PM, Sanderman R, Links TP, Schroevers MJ. Individual mindfulness-based cognitive therapy and cognitive behavior therapy for treating depressive symptoms in patients with diabetes: results of a randomized controlled trial. Diabetes Care. 2014 Sep;37(9):2427-34. doi: 10.2337/dc13-2918. Epub 2014 Jun 4. PMID 24898301
- [Background] Chiesa A, Serretti A. Mindfulness based cognitive therapy for psychiatric disorders: a systematic review and meta-analysis. Psychiatry Res. 2011 May 30;187(3):441-53. doi: 10.1016/j.psychres.2010.08.011. Epub 2010 Sep 16. PMID 20846726
- [Background] Goldberg SB, Tucker RP, Greene PA, Davidson RJ, Kearney DJ, Simpson TL. Mindfulness-based cognitive therapy for the treatment of current depressive symptoms: a meta-analysis. Cogn Behav Ther. 2019 Nov;48(6):445-462. doi: 10.1080/16506073.2018.1556330. Epub 2019 Feb 8. PMID 30732534